CLINICAL TRIAL: NCT05088330
Title: A Prospective Study of Daratumumab Combined With VRD in the Treatment of Patients With Newly Diagnosed Standard-risk Multiple Myeloma : a Single-center, Single-arm Clinical Study
Brief Title: A Study to Access of Daratumumab Combined With VRD in the Treatment of Patients With Standard-risk Newly Diagnosed MM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Fu chengcheng PhD, Principal Investigator, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-VRD-MM05
Record Dates: First submitted 2021-09-11; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Newly Diagnosed Multiple Myeloma
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: D-VRD
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- D-VRD (Experimental): treatment with D-VRD in NDMM
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — treatment with D-VRD in NDMM
  Other Names: DARA

SUMMARY:
This is an open-label, single arm study to access the effect of treatment with D-VRD in patients with newly diagnosed standard risk multiple myeloma.

DETAILED DESCRIPTION:
Research object:Newly diagnosed standard-risk multiple myeloma (NDMM) diagnosed according to the International Myeloma Working Group (IMWG) standards and who have been assessed to receive Autologous Stem Cell Transplantation (ASCT) but actively refused.Objective: To explore the therapeutic options of daratumamab (D) combined with bortezomib (V), lenalidomide (R) and dexamethasone ( d) for objective assessment of patients who can receive ASCT but not to receive transplantation.Main indicators:negative rate of minimal residual disease (MRD) upon completion of cycle 8 (24 weeks).

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years and ≤ 70 years, male or female；
2. Newly diagnosed multiple myeloma (NDMM) ；
3. Transplant-eligible；
4. Non-17p-, t(4;14) , t(14;16)；
5. Expected survival ≥12 weeks;
6. Eastern Cooperative Oncology Group (ECOG) scores 0 - 2.
7. Subjects should have adequate hemostatic and liver and kidney meet the following examination criteria: (without ongoing supportive treatments):

   1. Complete blood count (CBC) results: absolute neutrophil count（ANC） ≥ 1.0 × 109/L, platelet count ≥ 75 × 109/L (if the proportion of plasma cells in the bone marrow is > 50%, subjects with platelets ≥ 50 × 109/L will be eligible), Hb ≥ 70 g/L.
   2. Blood biochemistry: creatinine clearance ≥ 30 mL/min, alanine aminotransferase (ALT) ≤ 2.5 × upper limit normal (ULN)，aspartate aminotransferase (AST) ≤ 2.5 × ULN, total bilirubin ≤ 1.5 × ULN. Serum calcium ≤14.0 mg/dL (≤3.5 mmol/L);
8. Normal cardiopulmonary function;
9. The patient agrees to join the clinical trial and signs an informed consent form.

Exclusion Criteria

1. Poor hypertension control;
2. Have received ASCT or anti-tumor systemic therapy;
3. Peripheral neuropathy or neuralgia of grade 2 or higher;
4. During pregnancy or lactation or planning to become pregnant;
5. History of other malignant tumors within 5 years;
6. Subjects positive for any following tests: human immunodeficiency virus (HIV) antibody, Treponema pallidum (syphilis) antibody, hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) and HBV DNA.
7. Participating in other clinical trials;
8. Allergic to the drugs in the treatment plan;
9. Receiving any other experimental drugs or experimental medical devices;
10. The investigator believes that the patient has other conditions that are not suitable for participating in this study.
11. Patients with R-ISS Phase III

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of minimal residual disease negativity | end of 8 cycles
  rate of minimal residual disease negativity